CLINICAL TRIAL: NCT05192473
Title: A Prospective, Single-Arm, Multicenter, Feasibility Study to Evaluate Safety and Performance of the Amplitude Vascular System (AVS) Pulse Peripheral Intravascular Lithotripsy (IVL) for Treating Subjects With Calcific Femoropopliteal Arteries in Conjunction With Adjunctive Therapy
Brief Title: POWER: Pulse Intravascular Lithotripsy (Pulse IVL) to Open Vessels With Calcific Walls and Enhance Vascular Compliance and Remodeling
Acronym: POWER-PAD-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amplitude Vascular Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPF-001
Record Dates: First submitted 2021-12-09; First posted 2022-01-14 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lithotripsy Treatment (Experimental): Pulse Intravascular Lithotripsy System
  Device: Pulse Intravascular Lithotripsy Catheter
  Interventions: Device: Pulse Intravascular Lithotripsy System

INTERVENTIONS:
Device: Pulse Intravascular Lithotripsy System — Treatment with Pulse Intravascular Lithotripsy System

SUMMARY:
The POWER-PAD-1 Study is a first-in-human evaluation of the safety and performance of the Pulse Peripheral Intravascular Lithotripsy (IVL) Balloon Catheter to enroll up to twenty (20) subjects.

DETAILED DESCRIPTION:
Amplitude Vascular System intendeds to conduct a first-in-human evaluation of the safety and performance of the Pulse Peripheral Intravascular Lithotripsy (IVL) Balloon Catheter in subjects with stenotic lesions of the superficial femoral and/or popliteal arteries (Rutherford Category 2 to 4 of the target limb) with a reference vessel diameter (RVD) of 4mm to 6mm and a total length of <60mm. Up to twenty subjects will be enrolled and treated with the Pulse IVL lithotripsy and followed for 6 months. The Pulse Intravascular Lithotripsy Catheter is intended for the pulsatile lithotripsy-enhanced balloon dilation of lesions, including calcified and fibro-calcific lesions in the peripheral vasculature, such as the superficial femoral and popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years.
2. Subject is able and willing to comply with all assessments in the study.
3. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate, and has signed the approved consent form approved by the local Ethics Committee.
4. Rutherford clinical category 2, 3, or 4 of the target limb.
5. Resting ankle-brachial index (ABI) of ≤0.90, or ≤0.75 after exercise, of the target leg.
6. Moderate to severe calcification of target lesion(s) per pre-procedure CT scan. (Calcification must be: ≥180 degrees circumferential at some point in the lesion AND extend ≥50% length of lesion or absolute length ≥20mm.)
7. Flow-limiting target lesion reference vessel diameter is between 4.0mm and 6.5mm as determined by investigator
8. Target lesion length is ≤150mm
9. Subject life expectancy >1 year
10. Subject is intended to undergo angiographic and endovascular intervention in the opinion of the investigator(s) and/or per hospital protocols.
11. Subject agrees to undergo treatment with Pulse Peripheral Intravascular Lithotripsy.

Exclusion Criteria:

1. Rutherford Category 0, 1, 5, and 6.
2. Subject has active infection in the target leg requiring antibiotic therapy.
3. Planned major amputation of the target leg (transmetatarsal or higher).
4. In-stent restenosis within the target lesion(s).
5. Significant target vessel tortuosity (bends >30 degrees over the arc length of the balloon) or other parameters prohibiting access to the target lesion.
6. Chronic total occlusion of the target lesion(s) > 40mm.
7. Target lesion(s) within native or synthetic vessel grafts.
8. Chronic total occlusion of inflow vessel.
9. Lesion in contralateral limb requiring intervention within the next 30 days.
10. Subject has had any major (e.g., cardiac, peripheral, abdominal) surgical procedure or intervention unrelated to this study within 30 days prior to the index procedure or has planned major surgical procedure or intervention within 30 days of the index procedure.
11. Subject has significant stenosis (>50% stenosis) or occlusion of inflow tract (upstream disease) not successfully treated with percutaneous transluminal angioplasty (PTA) or percutaneous stent.
12. Deep heel ulcers or any evidence of osteomyelitis.
13. Subject requires treatment of a peripheral lesion on the ipsilateral limb distal to the target lesion(s) at the time of the enrollment / index procedure.
14. Subject has a known coagulopathy or has a bleeding diathesis, thrombocytopenia with platelet counts <100,000/microliter, or international normalized ratio >1.5.
15. Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
16. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
17. Subject has known allergy to urethane, nylon, or silicone.
18. Myocardial infarction within 60 days prior to enrollment.
19. History of stroke within 60 days prior to enrollment.
20. Subjects that are non-ambulatory and confined to bed.
21. Subject has life expectancy <12 months.
22. History of unstable coronary artery disease or other uncontrollable comorbidity resulting in hospitalization within the last 60 days prior to enrollment.
23. History of thrombolytic therapy within 2 weeks of enrollment.
24. Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 µmol/L or is on dialysis).
25. Women who are pregnant, breast-feeding, or intend to become pregnant
26. Subject is participating in another investigational drug, biological, or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints of this study, or subject is planning to participate in such studies prior to the completion of this study.
27. Subject has any other condition that, at the discretion of the Investigator, would preclude them completing the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Success | up to 24 hours
  Defined as successful delivery, balloon inflation, deflation, and retrieval of the intact study device without bust below rated burst pressure
Technical Success | up to 24 hours
  Defined as successful vascular access, completion of endovascular procedure with or without adjunctive therapy, and immediate achievement of less than or equal to 50% residual stenosis of the treated lesion on completion of angiography.
Procedural Success | up to 24 hours
  Defined as Device Success or Technical Success and absence of procedural complications
Major Adverse Events | 30 days
  A composite of either unplanned major amputation (above the ankle) or major reintervention of target limb defined as new unplanned surgical bypass graft, the use of thrombectomy or thrombolysis, major surgical graft revision such as a jump graft or an interposition graft, or bail-out stenting at 30 days.

SECONDARY OUTCOMES:
Freedom from target limb revascularization | 30 days and 6 months
  Freedom from clinically driven target lesion revascularization at 30-days and 6-months
Clinical Success | up to 24 hours
  Achievement of residual stenosis of the treated lesion on completion of angiography with or without adjunctive therapy
Rutherford Clinical Category | 6 months
  Improvement in Rutherford Class score at 6 months
Ankle-Brachial Index | 30 days
  Change in Ankle Brachial Index (ABI) of the target limb at 30 days
Quality of Life at 30 days and 6 months | 30 days and 6 months
  Assessed by EUROQOL - EQ-5D-5L descriptive system (Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression) questionnaire at 30 days and 6 months reported as a change from baseline.
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems
Walking Capacity | 30 days and 6 months
  Assessed by the Walking Impairment Questionnaire (WIQ) at 30 days and 6 months reported as a change from baseline.
VacuQol | 30 days and 6 months
  Change in VascuQol score from pre-procedure to 30-days and 6-months
Major Adverse Event | 30 days
  Major Adverse Limb event or procedure-related death at 30-days
Major Unplanned Amputation | 6 months
  Major Unplanned Amputation of the target limb at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital; Nelson Encanacion, MD, Principal Investigator — Centro Medico Moderno; Bibombe P Mwipatayi, MD, Principal Investigator — Royal Perth Hospital
Locations (3):
- Royal Perth Hospital, Perth, Western Australia, Australia
- Centro Medico Moderno, Santo Domingo, Dominican Republic
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No